CLINICAL TRIAL: NCT01734837
Title: Prospective Multicenter Observational Study (Registry) on the Aesculap DS Titanium Ligation Clips for Appendiceal Stump Closure.
Brief Title: TICAP - Titanium Clips for Appendiceal Stump Closure
Acronym: TICAP
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: Aesculap, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1111
Record Dates: First submitted 2012-10-25; First posted 2012-11-28 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Appendicitis
Keywords: Laparoscopic appendectomy; appendical stump closure
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: DS-Ligature Clip

SUMMARY:
Laparoscopic appendectomy is progressively accepted as the treatment of choice for acute appendicitis. Although the surgical technique of laparoscopic appendectomy has been well established, some controversy exists regarding the closure of the appendiceal stump. The available methods for stump closure are currently: pre-knotted loops (Roeder Loops or Endoloop, linear stapler and polymeric clips. A new device is a the DS Titanium Ligation Clip. The design of the DS-Clip is characterized by two parallel shanks.

The aim of this study is to collect data of a large number of patients treated with the product in real-life clinical routine.

ELIGIBILITY:
Inclusion:

* indication for a laparoscopic appendectomy
* informed consent

Inclusion criteria to be checked intraoperatively:

* conventional laparoscopic approach (no SILS, NOTES, SPA)
* Aesculap DS Titanium Ligation Clips were used

Exclusion:

* patient age under 16 years
* appendix is severely inflamed with involvement of the caecum

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult patients and children
Sampling Method: Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Applicability/feasibility of the DS Clips | 30 days after surgery
  Documentation of the number of successful (= completed stump closure) versus non-successful (= clip could not be applied) applications of the DS-Clip

SECONDARY OUTCOMES:
Intra- and post-operative complications related to surgery | 30 days after surgery
Duration of operation | intra-operative
Conversion rate to open surgery | 30 days
Length of hospitalization | 30 days

CONTACTS AND LOCATIONS:
Locations (9):
- United States (2):
  - Marina del Rey Hospital, Marina del Rey, California
  - St. Luke's University Hospital, Bethlehem, Pennsylvania
- Germany (7):
  - Vivantes Humboldt-Klinikum, Berlin
  - DRK Krankenhaus Clementinen, Hanover
  - University of Mainz, Department of Surgery, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum Memmingen, Memmingen
  - Katharinenhospital, Stuttgart
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen

REFERENCES:
- [Result] Rickert A, Kruger CM, Runkel N, Kuthe A, Koninger J, Jansen-Winkeln B, Gutt CN, Marcus DR, Hoey B, Wente MN, Kienle P. The TICAP-Study (titanium clips for appendicular stump closure): A prospective multicentre observational study on appendicular stump closure with an innovative titanium clip. BMC Surg. 2015 Jul 17;15:85. doi: 10.1186/s12893-015-0068-3. PMID 26185103